CLINICAL TRIAL: NCT04206306
Title: Functional Recovery Over the First Year After ICU Discharge：How ICU-delirium and ICU-acquired Weakness Interact
Brief Title: Functional Recovery Over the First Year After ICU Discharge
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201802070RIND
Record Dates: First submitted 2018-08-08; First posted 2019-12-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2021-07

CONDITIONS: Adult Patients; Intensive Care Unit
Keywords: Intensive Care Unit Acquired Delirium; Intensive Care Unit Survivor; Intensive Care Unit Acquired Weakness; Functional recovery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intensive Care Unit Acquired Delirium (ICU-AD) and Intensive Care Unit Acquired Weakness (ICU-AW) are common in critically ill, mechanically ventilated adult patients. As more patients survive ICU stays but suffer from long-term functional declines leading to unemployment and disability, research is urgently needed. The aims of this study are to: 1) describe the trajectory of physical functions one year after ICU discharge, including distance walked in 6 minutes (6MWD), hand grip (HGS), maximum inspiratory pressure (MIP), cognitive function (mini mental state examination,MMSE), physical function ICU test score (PFITs) , medical reserach council scale (MRC), medical research council questionnaire (MRC-Q)and basic and instrumental activities of daily living (ADL/IADL); 2) examine the incidences of ICU-AD and ICU-AW; and 3) test the interaction between ICU-AD and ICU-AW on one-year functional trajectories in the ICU survivors.4) compare two tools, the intensive care delirium screening checklist (ICDSC) and confusion assessment method for the ICU (CAM-ICU), for their predictive validity for outcomes related to delirium, hospital mortality and length of stay (LOS), and examined whether the tools' predictive validity was affected by patients' arousal status (RASS≥0, RASS<0).

DETAILED DESCRIPTION:
For this 3-year cohort study, consecutive ICU stay over 24 hours and adult patients (≧20 years) will be screened for enrollment at 6 medical ICUs in the National Taiwan University Hospital. Participants will be assessed daily for delirium occurrence for up to 14 days of ICU stay, and again upon ICU discharge. The instrument used for delirium are the confusion assessment method for ICU (CAM-ICU) and the intensive care delirium screening checklist (ICDSC). The 7 point rating scale of CAM-ICU-7 will also be used to rate the severity of delirium. Delirium assessment is possible,if the the patient's Richmond Agitation and Sedation Scale (RASS, -5~+4) is ≧ -3, -4~-5 are deeper levels of sedation (unarousable or responsive to painful stimulation only) cannot be assessed accurately. The CAM-ICU comprises four features which assess the following: acute change or fluctuation in mental status (Feature 1), inattention (Feature 2), disorganized thinking (Feature 3) or an altered level of consciousness (Feature 4). Patients are considered to have delirium if they present with both the first (acute onset and fluctuating course) and second (inattention) core symptoms and either the third (altered consciousness) or fourth (disorganized thinking) symptom. The ICDSC comprises eight items (score 0-8), ICDSC score of 4 or higher are considered delirium.

At ICU discharge,assess ICU-AW using a standardized protocol. Participants will be followed for one year after ICU discharge at 1, 3, 6, 12 months. A comprehensive functional evaluation (6-minute walking test, grip strength test, maximum inspiratory pressure test, mini-mental state exam, physical function ICU test score and basic and instrument activities of daily living questionnaires, medical research council scale and medical research council questionnaire) will be completed. Estimated 158 participants will be enrolled and followed for one year.

Data will be analyzed using the SPSS package. For example, the Generalized Estimating Equation (GEE) will be performed to delineate the trajectory of physical functions one year after ICU discharge and to test the interaction among ICU-AD, ICU-AW, and one-year functional trajectories. The findings will add to the development of intervention program to reduce ICU-AD and ICU-AW, thus promoting functional recovery for ICU survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is 20 years or older.

Exclusion Criteria:

* patients who presented with preexisting delirium at ICU admission
* patients who were placed on contact and droplet precaution
* patient who is long-term bedridden, moderate to severe dementia
* expected ICU length of stay less than 24 hours
* unable to communicate in Mandarin or Taiwanese
* unable to follow command completely

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive about patients (≧20 years) admitted to the six medical intensive care units at the National Taiwan University Hospital (NTUH).
Sampling Method: Non-Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2018-08-14 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline 6-min walking distance to one year after ICU discharge | Baseline at ICU discharge one month. One,two, three,six month and one year after ICU discharge
  Measured by distance walked in 6 minutes(6MWT) in meter
Change from baseline hand grip strength to one year after ICU discharge | Baseline at ICU discharge. One, two, three,six month and one year after ICU discharge
  Measured by hand grip strength (HGS) in kg, range from 20 to 65 kg, higher value indicated better musculoskeletal function
Maximum inspiratory pressure, from baseline to one year after ICU discharge | Baseline at ICU discharge one month. Two, three, six month and one year after ICU discharge
  Measured by maximum inspiratory pressure (MIP test ) in cmH2O, normal range < -20 cmH2O, lower value indicated better respiratory muscle condition
Change from baseline Mini-Mental State Examination to one year after ICU discharge | Baseline at ICU discharge. One, two, three, six month and one year after ICU discharge
  Measured by Mini-Mental State Examination (MMSE) in score, range from 0 to 30 score, higher score indicated better cognitive function
Physical function | Three months after ICU discharge
  Measured by Physical function ICU test score (PFITs)
Activities of daily living score, from baseline to one year after ICU discharge | Baseline before hospital admission. ICU discharge, one, two, three,six month and one year after ICU discharge
  Measured by basic activities of daily living (ADL) in score, range from 0-100 score, higher score indicated health condition
Instrumental activities of daily living score, from baseline to one year after ICU discharge | Baseline at ICU discharge one month. Two, three, six month and one year after ICU discharge
  Measured by instrumental activities of daily living (IADL) in score, range from 0 to 8 score, higher score indicated better health condition
Scores of Medical Research Council (MRC) scale, from baseline to one year after ICU discharge | Baseline at ICU discharge. One year after ICU discharge
  Measured by medical research council scale (MRC) in score, range from 0 to 60 score, higher score indicated better muscle strength
Self-report MRC questionnaire score | At ICU discharge one month
  range from 0 to 60, score greater than or equal to 48, classified as no muscle weakness
Sit-to-stand ability (yes/no) | Three months after ICU discharge
  Asking participants to rise from a seated position, with full body weight on the chair, to a standing posture, with their legs fully extended.

SECONDARY OUTCOMES:
ICU, hospital, and one-year mortality | death (yes/no) at ICU, at hospital, and one year after ICU discharge obtained by family interview and medical record
  death (yes/no) at ICU, at hospital, and one year after ICU discharge obtained by family interview and medical record
Length of ICU and hospital stay (day) | calculated a duration of ICU and hospitalization, obtained by medical record
  calculated a duration of ICU and hospitalization, obtained by medical record

OTHER OUTCOMES:
Time spent administering delirium tools | time spent (minutes) administering ICDSC vs CAM-ICU was automatically recorded by the REDCap data collection system
  time spent (minutes) administering ICDSC vs CAM-ICU was automatically recorded by the REDCap data collection system
Diagnostic accuracy of HGS and MIP as surrogate markers for ICU-AW | Baseline at ICU discharge
  Measured by the area under the ROC curve (AUC), sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV).

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Chia-Hui Chen Chen, PhD, Principal Investigator — School of Nursing, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Siao SF, Zheng YY, Wei YC, Boehm LM, Chen CC. Delirium and Weakness Acquired in the Intensive Care Unit: Individual and Combined Effects on 90-Day Mortality in Survivors of Critical Illness. J Clin Nurs. 2025 Sep;34(9):3620-3627. doi: 10.1111/jocn.17517. Epub 2024 Oct 29. PMID 39468861